CLINICAL TRIAL: NCT00568178
Title: A Randomized, Double-Blind, Parallel, Placebo or Amlodipine-Controlled Study of the Effects of Losartan on Proteinuria in Pediatric Patients With or Without Hypertension
Brief Title: An Extension Study Designed to Assess Effects of Losartan on Proteinuria in Pediatric Populations (MK-0954-326 AM1,EXT1(AM2))
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0954-326; 2006-006415-74 (EudraCT Number)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2009-10-30 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Losartan; Amlodipine; Enalapril; Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Losartan Double-Blind Base Study (12-weeks) (Experimental): Normotensive participants received losartan.
  Hypertensive participants received either active losartan (plus amlodipine placebo) OR active amlodipine (plus losartan placebo).
  Interventions: Drug: Losartan Potassium; Other: Comparator: Placebo (Losartan)
- Amlodipine Double-Blind Base Study (12-weeks) (Active Comparator): Hypertensive participants were randomized to receive either active losartan (plus amlodipine placebo) OR active amlodipine (plus losartan placebo) for 12 weeks.
  Interventions: Other: Comparator: Placebo (Losartan); Drug: Comparator: amlodipine besylate; Other: Comparator: Placebo (amlodipine besylate); Other: Placebo (Losartan)
- Losartan Open-Label Extension Phase (Month 36) (Experimental): Participants were were carried over from the base study into the long-term safety extension. Participants in the extension were randomly assigned to either losartan or enalapril regardless of their previous randomized treatment. Dosing during the extension period (i.e. starting dose and any titration) was up to the investigator and varied by patient).
  Interventions: Drug: Losartan Potassium
- Enalapril Open-Label Extension Phase (Month 36) (Active Comparator): Participants were were carried over from the base study into the long-term safety extension. Participants in the extension were randomly assigned to either losartan or enalapril regardless of their previous randomized treatment. Dosing during the extension period (i.e. starting dose and any titration) was up to the investigator and varied by patient).
  Interventions: Drug: Enalapril Maleate

INTERVENTIONS:
Drug: Losartan Potassium — Losartan Use During the Double-Blind Treatment Phase:
  Losartan potassium was administered orally as tablets; 25 or 50 milligrams (mg); or as a liquid suspension 2.5 mg/mL prepared for participants who weighed less than 25 kilograms (kg) or for those participants unable to swallow tablets. During the double-blind period, participants were initially randomized to either a once-daily weight-dependent dose of approximately 0.7 mg/kg (25 mg tablet; up to 50 mg per day) and at 2-weeks the dose was increased to a once-daily maximum weight-dependent dose of 1.4 mg/kg. The maximum dose of losartan, as specified in the protocol, was 50 mg/day (if the patient weighed <50 kg)
  or 100 mg/day (if the patient weighed ≥50 kg).
  Losartan Use During the Treatment Extension Phase:
  Dose modifications of the drug were left up to the discretion of the Investigators based on each participant's level of tolerance.
  Other Names: Cozaar®
  Arms: Losartan Double-Blind Base Study (12-weeks); Losartan Open-Label Extension Phase (Month 36)
Other: Comparator: Placebo (Losartan) — Placebo (losartan suspension), administered orally, once daily for 12 weeks
  Arms: Amlodipine Double-Blind Base Study (12-weeks); Losartan Double-Blind Base Study (12-weeks)
Drug: Comparator: amlodipine besylate — Amlodipine besylate (1 mg/mL) liquid suspension, oral administration, titrated to 0.2 mg/kg/day (5 mg maximum dose) per day for 12 Weeks
  Other Names: NORVASC®
  Arms: Amlodipine Double-Blind Base Study (12-weeks)
Other: Comparator: Placebo (amlodipine besylate) — Liquid suspension, 1mg/mL, titrated to 0.2 mg/kg/day (5 mg maximum dose) once daily, for 12 weeks
  Other Names: NORVASC®
  Arms: Amlodipine Double-Blind Base Study (12-weeks)
Other: Placebo (Losartan) — Normotensive patients randomized to losartan placebo for 12 weeks.
  Arms: Amlodipine Double-Blind Base Study (12-weeks)
Drug: Enalapril Maleate — Enalapril 2.5-, 5-, 10-, and 20-mg tablets or enalapril suspension (1 mg/mL), oral administration, once daily for 36 months.
  Other Names: Vasotec®; Renitec®
  Arms: Enalapril Open-Label Extension Phase (Month 36)

SUMMARY:
The purpose of this study is to evaluate the effects of losartan on proteinuria in pediatric patients.

DETAILED DESCRIPTION:
The study included a 12-week double-blind treatment phase and a 36-month open-label extension phase. Participants who completed or discontinued the initial 12-week phase of the study and who opted to participate in the open label extension phase were randomized to either losartan or enalapril at a dose of the investigator's choosing for the duration of the extension. The open label extension was designed to continue until the 100th participant completed 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 1 to 17 years of age
* Able to provide a first-morning urine sample each day during the study
* Documented history of proteinuria associated with chronic kidney disease of any origin
* Signed consent of parent and/or legal guardian

Exclusion Criteria:

* Pregnant and/or nursing
* Requires more than 2 medications to control high blood pressure
* Has undergone major organ transplantation (e.g. heart, kidney, liver)
* Known sensitivity to losartan or other similar drugs, or any history of angioneurotic edema
* Known sensitivity to amlodipine or other calcium channel blocker
* Requires cyclosporine to treat renal disease (kidney disease)

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Webb NJ, Shahinfar S, Wells TG, Massaad R, Gleim GW, McCrary Sisk C, Lam C. Losartan and enalapril are comparable in reducing proteinuria in children with Alport syndrome. Pediatr Nephrol. 2013 May;28(5):737-43. doi: 10.1007/s00467-012-2372-9. Epub 2012 Dec 4. PMID 23207876
- [Derived] Webb NJ, Shahinfar S, Wells TG, Massaad R, Gleim GW, Santoro EP, Sisk CM, Lam C. Losartan and enalapril are comparable in reducing proteinuria in children. Kidney Int. 2012 Oct;82(7):819-26. doi: 10.1038/ki.2012.210. Epub 2012 Jun 27. PMID 22739977
- [Derived] Webb NJ, Lam C, Shahinfar S, Strehlau J, Wells TG, Gleim GW, Le Bailly De Tilleghem C. Efficacy and safety of losartan in children with Alport syndrome--results from a subgroup analysis of a prospective, randomized, placebo- or amlodipine-controlled trial. Nephrol Dial Transplant. 2011 Aug;26(8):2521-6. doi: 10.1093/ndt/gfq797. Epub 2011 Feb 1. PMID 21285125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of March 2011, the study was completed.
  Phase III First Patient In: 21Jun07; Last Patient Last Visit (double-blind base study): 16Sep08; and (open-label extension): 31Mar11. The study included 52 centers (USA, Europe, Latin America, and Asia) and participants included children aged 6-17 (hypertensive) or 1-17 (normotensive) with proteinuria.
Pre-assignment Details: During a 4-week, single-blind run-in participants received losartan placebo (normotensive) or amlodipine (hypertensive) and underwent wash-out of anti-hypertensive agents. To qualify for randomization, participants had to have a mean urine Pr/Cr ratio of ≥0.3 gram/gram (gm/gm) derived from baseline urine samples.
Groups:
- Losartan Double Blind Normortensive: Normotensive participants who were randomized to losartan.
  Losartan dispensed as tablets or suspension depending on participant weight and ability to swallow tablets.
  Losartan suspension dosing: 0.7 milligram/kilograms/day (mg/kg/day) titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks. Losartan tablet dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks; or losartan placebo.
- Placebo Double Blind Normotensive: Normotensive participants who were randomized to losartan placebo.
  Losartan placebo dispensed as tablets or suspension depending on participant weight and ability to swallow tablets.
  Losartan placebo suspension dosing: 0.7 mg/kg/day titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks.
  Losartan placebo tablet dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks.
- Losartan Double Blind Hypertensive: Hypertensive patients who were randomized to receive losartan and amlodipine placebo for 12 weeks.
  Losartan dispensed as tablets or suspension depending on participant weight and ability to swallow tablets. Amlodipine placebo dispensed as suspension for duration of study.
  Losartan suspension dosing: 0.7 milligram/kilograms/day (mg/kg/day) titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks. Amlodipine placebo suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan tablet dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks.
- Amlodipine Double Blind Hypertensive: Hypertensive patients who were randomized to receive amlodipine and losartan placebo for 12 weeks.
  Losartan placebo dispensed as tablets or suspension depending on participant weight and ability to swallow tablets.
  Losartan placebo suspension dosing: 0.7 mg/kg/day titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks.
  Amlodipine suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan placebo tablet dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks.
- Losartan Open Label Extension: Participants were stratified based on assigned treatment in the double-blind treatment phase and were randomized in a 1:1 ratio to either losartan or enalapril.
  Dosing of study medication during the extension phase of the study was at the investigator's discretion.
  Losartan 25-mg and 50-mg tablets were available for patients able to swallow tablets. For patients unable to swallow tablets, or who weighed <25 kg, losartan suspension (2.5 mg/ml) was prepared.
- Enalapril Open Label Extension: Participants were stratified based on assigned treatment in the double-blind treatment phase and were randomized in a 1:1 ratio to either losartan or enalapril.
  Dosing of study medication during the extension phase of the study was at the investigator's discretion.
  Enalapril 2.5-, 5-, 10-, and 20-mg tablets were available for participants able to swallow tablets. For participants unable to swallow tablets, or who weighed <25 kg, enalapril suspension (1 mg/mL) was prepared.
Period: Double Blind Base Study
Arm/Group | Losartan Double Blind Normortensive | Placebo Double Blind Normotensive | Losartan Double Blind Hypertensive | Amlodipine Double Blind Hypertensive | Losartan Open Label Extension | Enalapril Open Label Extension
Started | 122 | 124 | 30 | 30 | 0 | 0
Completed | 116 | 118 | 29 | 25 | 0 | 0
Not Completed | 6 | 6 | 1 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 0 | 0
Period: Open Label Extension
Arm/Group | Losartan Double Blind Normortensive | Placebo Double Blind Normotensive | Losartan Double Blind Hypertensive | Amlodipine Double Blind Hypertensive | Losartan Open Label Extension | Enalapril Open Label Extension
Started | 0 | 0 | 0 | 0 | 134 | 134
Completed | 0 | 0 | 0 | 0 | 55 | 54
Not Completed | 0 | 0 | 0 | 0 | 79 | 80
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 11 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6 | 11
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 9 | 8
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Termination of Trial | 0 | 0 | 0 | 0 | 45 | 47
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Losartan: Four arms combined to 2 groups (losartan & amlodipine/placebo) for reporting and compared those who took losartan to those who did not (i.e., participants took amlodipine and/or placebo).
  "Losartan" group: Normotensives were randomized to losartan and Hypertensives were randomized to losartan & amlodipine placebo.
  Losartan dispensed as tablets or suspension depending on patient weight and ability to swallow tablets. Amlodipine placebo dispensed as suspension for duration of study.
  Losartan suspension dosing: 0.7 milligram/kilograms/day (mg/kg/day) titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks. Amlodipine placebo suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks.
- Amlodipine/Placebo: "Amlodipine/Placebo" group includes the following: Normotensive patients randomized to losartan. Hypertensive patients randomized to amlodipine and losartan placebo.
  Losartan placebo dispensed as tablets or suspension depending on patient weight and ability to swallow tablets. Amlodipine dispensed as suspension for duration of study. Losartan placebo suspension dosing: 0.7 mg/kg/day titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks.
  Amlodipine suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan placebo tablet dosing: 25 mg/day orally titrated to 50 mg/day (patients <50 kg) OR 50 mg/day orally titrated to 100 mg/day (patients ≥50 kg) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Losartan | Amlodipine/Placebo | Total
Number analyzed (Participants) | 152 | 154 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.7) | 9.7 (4.6) | 10.1 (4.7)
Age, Customized [Number; unit: participants]
  ≤6 Years of Age | 33 | 42 | 75
  7-12 Years of Age | 57 | 57 | 114
  13-17 Years of Age | 62 | 55 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 86 | 90 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 82 | 161
  Not Hispanic or Latino | 73 | 72 | 145
  Unknown or Not Reported | 0 | 0 | 0
Hypertensive [Number; unit: Participants] — Sitting systolic blood pressure (SiSBP) or diastolic blood pressure (SiDBP) ≥90th percentile AND participant on medication for proteinuria/hypertension OR SiSBP or SiDBP ≥95th percentile AND participant NOT on medication for proteinuria/hypertension OR documented hypertension and on anti-hypertensive medication, whether or not medicated for proteinuria.
  Participants
    Yes | 30 | 30 | 60
    No | 122 | 124 | 246
Prior Angiotensin Converting Enzyme Inhibitor /Angiotensin II Type I Receptor Blocker (ACE-I/ARB)Use [Number; unit: Participants]
  Yes | 83 | 81 | 164
  No | 69 | 73 | 142
Race [Number; unit: participants]
  Asian | 26 | 26 | 52
  Black | 5 | 5 | 10
  Multi-Racial | 36 | 34 | 70
  White | 77 | 85 | 162
  Other | 8 | 4 | 12
Region [Number; unit: Participants]
  United States | 15 | 10 | 25
  Outside of United States | 137 | 144 | 281
Tanner Stage [Number; unit: Participants] — A scale of physical development.
  The scale defines physical measurements of development based on external primary and secondary sex characteristics, such as the size of the breasts, genitalia, and development of pubic hair.
  Stages range from I to V with I being the least developed.
  Participants
    Stage I | 69 | 78 | 147
    Stage II | 26 | 21 | 47
    Stage III | 22 | 18 | 40
    Stage IV | 23 | 24 | 47
    Stage V | 12 | 13 | 25
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m2)] | 19.8 (5.5) | 19.2 (4.2) | 19.5 (4.9)
Duration of Hypertension [Mean (Standard Deviation); unit: Years] | 4.8 (4.1) | 6.1 (4.8) | 5.5 (4.5)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 135.8 (27.3) | 132.0 (28.4) | 133.9 (27.9)
Protein-to-Creatinine Ratio [Mean (Standard Deviation); unit: grams/grams] | 2.2 (2.6) | 2.8 (3.8) | 2.5 (3.3)
Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 66.8 (10.7) | 67.8 (11.6) | 67.3 (11.2)
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 106.0 (13.4) | 107.2 (13.8) | 106.6 (13.6)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 39.6 (21.0) | 36.4 (19.5) | 38.0 (20.3)

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Treatment Phase: Percent Change From Baseline in Urinary Protein/Creatinine (Pr/Cr) Ratio (gm/gm) at Week 12
Description: Change in urinary protein excretion, determined as urinary Pr/Cr ratio compared to baseline*, after approximately twelve weeks of treatment.
  Baseline is defined as values obtained at Visit 3, Week (-1) during the Single Blind Run-in period.
Time Frame: Baseline and Week 12
Population: Full Analysis Set included all randomized participants who took at least one dose of study drug and had baseline and post randomization measurements available
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change in Pr/Cr
Groups:
- Losartan: Participants were randomized in a 1:1 ratio within each stratum: hypertensive patients (6 to 17 years of age) were randomized to either amlodipine or losartan; normotensive patients (1 to 17 years of age) were randomized to either placebo or losartan. Losartan (or placebo) therapy was administered orally, in tablet or suspension form, at an initial dose of approximately 0.7 mg/kg once daily (up to 50 or 100 mg total daily dose, weight-dependent). Participants who were randomized to losartan were assigned to a normotensive or hypertensive group, based on clinical profile.
- Amlodipine/Placebo: "Amlodipine/Placebo" group includes the following: Normotensive patients randomized to losartan placebo. Hypertensive patients randomized to amlodipine and losartan placebo.
  Losartan placebo dispensed as tablets or suspension depending on patient weight and ability to swallow tablets. Amlodipine dispensed as suspension for duration of study. Losartan placebo suspension dosing: 0.7 mg/kg/day titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks.
  Amlodipine suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan placebo tablet dosing: 25 mg/day orally titrated to 50 mg/day (patients <50 kg) OR 50 mg/day orally titrated to 100 mg/day (patients ≥50 kg) for 12 weeks.
Arm/Group | Losartan | Amlodipine/Placebo
Number analyzed (Participants) | 150 | 152
Percent Change in Pr/Cr | -35.80 [-43.11 to -27.55] | 1.37 [-10.27 to 14.51]
Statistical Analysis 1: Comparison: Losartan vs Amlodipine/Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Ratio in Geometric Mean = 0.63, 95% CI 2-sided [0.54 to 0.74]

2. Secondary Outcome: Double-Blind Treatment Phase: Change From Baseline in Systolic Blood Pressure in Hypertensive Participants at Week 12
Time Frame: Baseline and Week 12
Population: All-Participants-As-Treated population which included all randomized participants who received at least 1 dose of study therapy, and each participant was counted in the treatment group of the drug they actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Losartan-Hypertensive Participants: Group includes hypertensive participants who were randomized to losartan and amlodipine placebo.
- Amlodipine-Hypertensive Participants: Group includes hypertensive participants who were randomized to amlodipine and losartan placebo.
Arm/Group | Losartan-Hypertensive Participants | Amlodipine-Hypertensive Participants
Number analyzed (Participants) | 30 | 30
mm Hg | -5.5 [-8.6 to -2.4] | -0.1 [-3.3 to 3.1]
Statistical Analysis 1: Comparison: Losartan-Hypertensive Participants vs Amlodipine-Hypertensive Participants; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -5.4, 95% CI [-9.9 to -1.0]

3. Secondary Outcome: Double-Blind Treatment Phase: Change From Baseline in Diastolic Blood Pressure in Hypertensive Participants at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Losartan-Hypertensive Participants | Amlodipine-Hypertensive Participants
Number analyzed (Participants) | 30 | 30
mm Hg | -3.8 [-7.0 to -0.7] | 0.8 [-2.5 to 4.1]
Statistical Analysis 1: Comparison: Losartan-Hypertensive Participants vs Amlodipine-Hypertensive Participants; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -4.6, 95% CI [-9.2 to -0.1]

4. Primary Outcome: Open Label Extension: Percent Change From Baseline of Urinary Pr/Cr Ratio (gm/gm) at Month 36
Description: Change in urinary protein excretion, determined as urinary Pr/Cr ratio compared to baseline*, after approximately three years of treatment.
  *The baseline for efficacy data in the extension was defined as the last value obtained in the double-blind treatment phase.
Time Frame: Baseline and Month 36
Population: Data for analysis was obtained only from participants who had: 1) Baseline measure of Pr/Cr, 2) At least one dose of study drug, and 3) Post randomization measure of Pr/Cr. The number of participants was determined by including only the individuals who satisfied the criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change in Pr/Cr
Groups:
- Losartan Open Label Extension; Enalapril Open Label Extension: All participants who completed the 12-week double-blind treatment phase (or discontinued early due to increased proteinuria) were invited to participate in the open-label extension. Participants were randomized in a 1:1 ratio to either losartan or enalapril therapy. The duration of the extension varied, depending on the time of enrollment. All participants who entered the extension could continue until the 100th participant completed approximately 3 years of follow-up.
Arm/Group | Losartan Open Label Extension | Enalapril Open Label Extension
Number analyzed (Participants) | 130 | 130
Percent Change in Pr/Cr | -30.01 (5.02) [-44.35 to -11.98] | -40.45 (2.10) [-52.45 to -25.42]
Statistical Analysis 1: Comparison: Losartan Open Label Extension vs Enalapril Open Label Extension; Test type: Superiority or Other; Mixed Models Analysis — No P Value was calculated for this outcome; An unstructured variance-covariance was used; Geometric Mean Ratio = 1.18, 95% CI 2-sided [0.86 to 1.60]

5. Primary Outcome: Open Label Extension: Change From Baseline in Glomerular Filtration Rate (GFR) at Month 36
Description: The outcome measure of glomerular filtration rate was based on mL/min/1.73m^2, as determined by the Schwartz formula:
  GFR = _____0.55 x height (cm)_______ divided by serum creatinine (mg/dL)
  GFR values were compared to the baseline GFR measure.
  [Note: For male participants, ages 13 to 17 years, 0.70 was used as
  the multiplier in place of 0.55]
  Baseline in regard to the extension is defined as the last value obtained in the double-blind treatment phase.
Time Frame: Baseline and Month 36
Population: Data for analysis was obtained only from participants who had: 1) Baseline measure of Pr/Cr, 2) At least one dose of study drug, and 3) Post randomization measure of Pr/Cr. The number of participants was determined by including only individuals who satisfied the criteria.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in GFR mL/min1.73m^2
Groups:
- Losartan Open Label Extension; Enalapril Open Label Extension: All participants who completed the 12-week double-blind treatment phase (or discontinued early due to increased proteinuria) were invited to participate in the open-label extension and were randomly assigned using a 1:1 ratio to either losartan or enalapril therapy. The duration of the extension varied, depending on the time of enrollment. All patients who entered the extension continued until the 100th patient completed approximately 3 years of follow-up.
Arm/Group | Losartan Open Label Extension | Enalapril Open Label Extension
Number analyzed (Participants) | 127 | 127
Change in GFR mL/min1.73m^2 | 3.3 (66.3) [-5.2 to 11.7] | 7.0 (53.2) [-1.4 to 15.4]
Statistical Analysis 1: Comparison: Losartan Open Label Extension vs Enalapril Open Label Extension; Test type: Superiority or Other; Mixed Models Analysis — A P-Value was not calculated for this outcome; Least Square Mean = -3.8, 95% CI [-15.2 to 7.6]

ADVERSE EVENTS:
Groups:
- Losartan: Double-Blind Base Study: Four arms combined to 2 groups (losartan & amlodipine/placebo) for reporting and compared those who took losartan to those who did not (i.e., participants took amlodipine and/or placebo).
  "Losartan" group: Normotensives were randomized to losartan and Hypertensives were randomized to losartan & amlodipine placebo.
  Losartan dispensed as tablets or suspension depending on patient weight and ability to swallow tablets. Amlodipine placebo dispensed as suspension for duration of study.
  Losartan suspension dosing: 0.7 milligram/kilograms/day (mg/kg/day) titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks. Amlodipine placebo suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan dosing: 25 mg/day orally titrated to 50 mg/day (participants <50 kg) OR 50 mg/day orally titrated to 100 mg/day (participants ≥50 kg) for 12 weeks.
- Amlodipine/Placebo: Double-Blind Base Study: "Amlodipine/Placebo" group includes the following: Normotensive patients randomized to losartan placebo. Hypertensive patients randomized to amlodipine and losartan placebo.
  Losartan placebo dispensed as tablets or suspension depending on patient weight and ability to swallow tablets. Amlodipine dispensed as suspension for duration of study. Losartan placebo suspension dosing: 0.7 mg/kg/day titrated at 2 weeks to 1.4 mg/kg/day orally (maximum 50 mg if <50 kg or 100 mg if ≥50 kg) for 12 weeks.
  Amlodipine suspension dosing: starting dose 0.05 or 0.1 titrated to 0.2 mg/kg/day orally (max 5 mg/day) after 2 weeks if necessary to control blood pressure for 12 weeks. Losartan placebo tablet dosing: 25 mg/day orally titrated to 50 mg/day (patients <50 kg) OR 50 mg/day orally titrated to 100 mg/day (patients ≥50 kg) for 12 weeks.
- Losartan Open-Label Extension: Please note that the open label participant population was derived exclusively from the original base study population. There was no additional recruitment.
  Participants were randomized to either losartan or enalapril, administered in an unblinded fashion (placebo was not used) for the duration of the study. The maximum dose of losartan was 50 mg/day (if the participant weighed <50 kg) or 100 mg/day (if the participant weighed ≥50 kg) Losartan 25-mg and 50-mg tablets were available for participants able to swallow tablets, and losartan suspension (2.5 mg/ml) was prepared for participants unable to swallow tablets, or for those who weighed <25 kg.
- Enalapril: Open-Label Extension: Please note that the open label participant population was derived exclusively from the original base study population. There was no additional recruitment.
  Participants were randomized to either losartan or enalapril, administered in an unblinded fashion (placebo was not used) for the duration of the study. The maximum specified dose of enalapril was 40 mg/day. For participants unable to swallow tablets, or for those who weighed <25 kg, enalapril suspension (1 mg/mL) was prepared. The starting dose of drug and any adjustments during the open-label period were at the discretion of the investigator.
Arm/Group | Losartan: Double-Blind Base Study | Amlodipine/Placebo: Double-Blind Base Study | Losartan Open-Label Extension | Enalapril: Open-Label Extension
Serious Adverse Events (participants affected / at risk) | 8/152 | 5/154 | 27/134 | 25/134
Other Adverse Events (participants affected / at risk) | 71/152 | 66/154 | 83/134 | 78/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan: Double-Blind Base Study (N=152) | Amlodipine/Placebo: Double-Blind Base Study (N=154) | Losartan Open-Label Extension (N=134) | Enalapril: Open-Label Extension (N=134)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipomeningocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somatoform disorder neurologic (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan: Double-Blind Base Study (N=152) | Amlodipine/Placebo: Double-Blind Base Study (N=154) | Losartan Open-Label Extension (N=134) | Enalapril: Open-Label Extension (N=134)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 11 (12) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 7 (7) | 12 (15) | 7 (9)
Vomiting (Gastrointestinal disorders) | 6 (8) | 4 (4) | 16 (22) | 4 (4)
Pyrexia (General disorders) | 6 (6) | 2 (2) | 8 (10) | 7 (9)
Bronchitis (Infections and infestations) | 9 (10) | 8 (8) | 9 (13) | 9 (10)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 9 (15) | 6 (10)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 3 (4) | 7 (9)
Nasopharyngitis (Infections and infestations) | 24 (28) | 19 (22) | 31 (40) | 20 (28)
Pharyngitis (Infections and infestations) | 6 (6) | 6 (7) | 21 (44) | 20 (31)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 8 (11) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 9 (13) | 15 (50) | 9 (20)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 10 (14) | 10 (15)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 8 (10) | 6 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5) | 9 (15)
Dizziness (Nervous system disorders) | 6 (6) | 3 (3) | 3 (3) | 7 (10)
Headache (Nervous system disorders) | 13 (24) | 20 (31) | 7 (19) | 12 (23)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 8 (9) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (8) | 8 (9) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.